CLINICAL TRIAL: NCT05725642
Title: Prevalence Study and Identification of Factors Prognosis of Obstructive Sleep Apnea Syndrome Sleep in Pregnant Women
Acronym: SAOSPRONOS
Status: Not yet recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00981-42
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Polysomnography — Polysomnography

SUMMARY:
The exact prevalence of sleep-disordered breathing in pregnant women is not known. The results of a analysis of a small cohort of 105 pregnant women adjusted to body mass index estimate a prevalence of 8.4% in first quarter and 19.7% in the third quarter.

In this context, this study proposes to assess the prevalence of sleep-disordered breathing in pregnant women of the Private Hospital of the Loire and to identify the risks associated with these disorders by systematically proposing a polysomnography.

DETAILED DESCRIPTION:
Pregnancy brings physical and hormonal changes and sleep is impaired by heartburn, cramps, frequent urination, fetal movements... Snoring is commonly observed in pregnant women at the end of the second and third trimester. Snoring can be a manifestation of OSAS. It has been shown that the apnea-hypopnea index (AHI) increases during pregnancy, at the third quarter. Physiological changes associated with pregnancy increase the risk of OSAS. In pregnant women, sleep deprivation leads to increased risk of gestational diabetes, high blood pressure, preeclampsia and antenatal depression, but also a risk of premature delivery or having a child with a delay in growth.

Finally, the exact prevalence of sleep-disordered breathing in pregnant women is not known. The results of a analysis of a small cohort of 105 pregnant women adjusted to body mass index estimate a prevalence of 8.4% in first quarter and 19.7% in the third quarter.

In this context, this study proposes to assess the prevalence of sleep-disordered breathing in pregnant women of the Private Hospital of the Loire and to identify the risks associated with these disorders by systematically proposing a polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman aged 18 and over.
* Pregnant woman who has not yet completed her consultation of the 1st quarter.
* Woman accepting the achievement of, at most, 2 polysomnographies.
* Affiliated participant or beneficiary of a security regime social.
* Participant having been informed of the study and not objecting to the use of her data.
* Authorization to collect and use the baby's data.

Exclusion Criteria:

* Participation in another clinical study.
* Participant with protected status: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Participant hospitalized without consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
OSAS Diagnosis with polysomnography | 9 months
  Diagnosis of OSAS with polysomnography, prior to the study, or during the first 2 trimesters of pregnancy

IPD SHARING:
Plan to Share IPD: No